CLINICAL TRIAL: NCT04436718
Title: Does Serial Ultrasonographic Assessment for Extravascular Lung Water and IVC Measurement Affect Outcomes in Inpatient Heart Failure Management?
Brief Title: Does Ultrasound Assessment for Extravascular Lung Water and IVC Measurement Affect Outcomes in Inpatient Heart Failure Management?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riverside University Health System Medical Center (Other)
Responsible Party: Principal Investigator, Michael Ulrich MD, Associate Medical Program Director, Riverside University Health System Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1374867-5
Record Dates: First submitted 2019-11-20; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Point of care ultrasound; Focused cardiac ultrasound; heart failure; inferior vena cava; POCUS; CHF; FCU; acute heart failure; decompensated heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized open label controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Daily POCUS (Experimental): Patients are assessed by facility experts with daily chest ultrasound and findings of interstitial syndrome and IVC measurement are reported to primary care providers.
  Interventions: Diagnostic Test: Daily pocus exam
- Usual care (No Intervention): Patients are assessed daily by primary care providers per usual care.

INTERVENTIONS:
Diagnostic Test: Daily pocus exam — Daily evaluation of lung ultrasound for B line artifacts plus IVC assessments
  Arms: Daily POCUS

SUMMARY:
This study evaluates daily POCUS/FCU exams on patients admitted for acute decompensated heart failure with primary end point of acute kidney injury while in hospital.

DETAILED DESCRIPTION:
Patients with admitted to hospital with Acute Decompensated Heart failure (ADHF) suffer a significant morbidity and premature mortality. Administration of intravenous (IV) diuretics is largely guided by clinical judgment based on physical exam, net fluid measurement, changes in daily weights and chest x-ray findings. The key objective is to promote adequate diuresis while improving symptoms, without compromising renal function. Laboratory tests demonstrating hemo-concentration, increasing BUN, and increasing creatinine have been proposed as positive prognostic indicators in patients receiving IV diuretic therapy but these methods suffer from inadequate predictive value. Observational studies have identified worsening renal failure (WRF) in patients admitted for heart failure as an important clinical entity associated with worsening clinical outcomes.

Point of care Ultrasound (POCUS) has the potential to fill an unmet need for monitoring patients recieving IV diuretic therapy. POCUS provides clinicians with immediate diagnostic information obtained and interpreted at bedside that can augment and enhance the physical examination. Numerous studies have examined POCUS assessment of pulmonary edema and measurement of the Inferior Vena Cava (IVC) to estimate hemodynamic parameters for patients with acute decompensated heart failure (ADHF). No study to date has examined POCUS effect on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 admitted for acute decompensated heart failure exacerbation as primary admission diagnosis from Emergency department to General Medicine ward that are administered diuretic therapy expected to be admitted for two days or more.

Exclusion Criteria:

1. Decline consent for study
2. If admitted and research team not available for consent and initial evaluation prior within 6 hours of first diuretic administration
3. Patients in whom diuretics will not be utilized (i.e. anuric, ESRD on HD)
4. Inability to assess IVC (surgical anatomy, body habitus, Ileus, etc.)
5. Patients admitted to ICU
6. Patients currently on positive pressure ventilation (BiPAP)
7. Patients discharged from the emergency department
8. Patients discharged prior to evaluation by the POCUS team

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Worsening renal failure | During hospitalization typically one week
  Serum Creatnine levels measured in mg/dL

SECONDARY OUTCOMES:
Length of stay | During hospitalization typically one week
  Measured in days from initial admission to discharge

CONTACTS AND LOCATIONS:
Locations (1):
- RUHS Medical center, Moreno Valley, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT04436718/Prot_000.pdf
  • Informed Consent Form (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT04436718/ICF_001.pdf